CLINICAL TRIAL: NCT05363098
Title: Investigating the Effects of Expiratory Flow Limitation and the Effects of Spontaneous Breathing on Intracranial Pressure. An Observational Clinical Study on Neurosurgical Patients.
Brief Title: The Cerebral-Respiratory Interaction During Spontaneous Breathing Ventilation in Neurosurgical Patients (CeRes-SB)
Acronym: CeRes-SB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Mariangela Pellegrini, Principal Investigator, Uppsala University
Other Study IDs: CeRes-SB
Record Dates: First submitted 2022-04-27; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Mechanical Ventilation Complication; Neurological Complication; Respiratory Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood gas analysis sampled daily shortly before respiratory mechanics data recording
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically ventilated neurosurgical patients: Observational study in mechanically ventilated neurosurgical patients
  Interventions: Other: Mechanically ventilated neurosurgical patients

INTERVENTIONS:
Other: Mechanically ventilated neurosurgical patients — Observational study where respiratory variables and intracranial pressure will be measured during assisted mechanical ventilation. No intervention is planned.

SUMMARY:
Mechanical ventilation (MV) is a life-saving supportive therapy and one of the most common interventions implemented in intensive care.

To date, only the inspiratory phase of breathing has been extensively investigated, and new MV methods have been implemented to reduce its harmful effects. Despite this, lung injury still occurs and propagates, causing multiorgan failure and patient deaths. The expiratory phase is considered unharmful and is not monitored or assisted during MV. In animal experiments, we recently showed that the loss of diaphragmatic contraction during expiration can harm the lungs during MV. During mechanical ventilation, the expiratory phase of breathing is completely disregarded. However, in all conditions that promote lung collapse, peripheral airways gradually compress and close throughout the expiration, potentially worsening lung injury.

This cyclical lung collapse and consequent air-trapping may have an impact on the Starling resistor mechanisms that regulate venous return from the brain, potentially affecting cerebral perfusion and intracranial pressure.

This study will investigate the incidence and the consequences of an uncontrolled expiration and expiratory lung collapse in spontaneously breathing critically ill neurosurgical patients during mechanical ventilation.

Electrical impedance tomography measurements , oesophagus and gastric pressure, electrical activity of the diaphragm and intracranial pressure will be acquired in a synchronised manner during controlled mechanical ventilation, on a daily bases during assisted mechanical ventilation.

ELIGIBILITY:
Neurosurgical patients on mechanical ventilation and with ongoing intracerebral pressure monitoring will be included in the study

Inclusion Criteria:

* Age >18 years;
* MV expected for more than 72 hours;
* Not pregnant;
* Informed consent from patient or next of kin.

Exclusion Criteria:

* Previously demonstrated paralysis of the diaphragm or know pathology of the phrenic nerve or neuromuscular disorder;
* Chest tube;
* Patients with clinical conditions that contraindicate the insertion of esophageal/gastric catheters (e.g., esophagus rupture, esophageal bleeding);
* Pacemaker and/or implantable cardioverter defibrillator, these last being a contraindication for EIT;
* Hemicraniectomy. In case of late hemicraniectomy (after patient inclusion), the patient will drop-out from the study.

Relative contraindication: in case of skull base fracture the patient can be included only if oesophageal/gastric and NAVA catheters can be inserted orally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients recruitment will be kept equally distributed between sexes.
Study Population: Critically ill adult patients affected by acute brain injury (e.g., subarachnoid hemorrhage, subdural hemorrhage, epidural hemorrhage, traumatic brain injury, intracerebral hemorrhage) admitted to the NICU of Uppsala. Consecutive patients will be prospectively screened for eligibility according to inclusion criteria
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of uncontrolled expiration | during the period of assisted mechanical ventilation, an average of 14 days
  The incidence of uncontrolled expiration and consequent expiratory lung collapse (determined by changes in expiratory flow and time constant) during assisted ventilation in neurosurgical patients.
Correlation between uncontrolled expiration and intracranial pressure | During the period of assisted mechanical ventilation, an average of 14 days
  The influence of an uncontrolled expiration (defined by expiratory flow, expiratory EAdi and thoracic impedance) on intracranial pressure in neurosurgical patients.

SECONDARY OUTCOMES:
Intensive care unit (ICU) and hospital length of stay (LOS) | At ICU/hospital discharge, an average of 30 days
  Correlation between lung collapse and LOS
Number of days of mechanical ventilation | At ICU discharge, an average of 20 days
  Correlation between lung collapse and days of mechanical ventilation
90-days mortality from intensive care unit admission | 90 days after hospital discharge
  Correlation between lung collapse and 90-days mortality
30-day and 90-days neurological and functional outcomes | 90 days after hospital discharge
  Correlation between lung collapse and 30-day and 90-days neurological and functional outcomes (Disability Rating Scale, clinical frailty score, Glasgow Outcome Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Pellegrini, MD, PhD, Principal Investigator — Uppsala University Hospital, Uppsala University

IPD SHARING:
Plan to Share IPD: No